CLINICAL TRIAL: NCT03995576
Title: Incidence of Inadvertent Intercostal or Epidural Spread During Thoracic Sympathetic Ganglion Block
Brief Title: Thoracic Sympathetic Ganglion Block Inadvertent Spread
Status: Completed | Type: Observational
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2019-05-028-004
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Thoracic; Sympathetic Ganglion, Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: thoracic sympathetic ganglion block — thoracic sympathetic ganglion block which needle reaches posterolateral vertebral body

SUMMARY:
This study wants to identify the incidence of inadvertend intercostal or epidural spread of thoracic sympathetic block

DETAILED DESCRIPTION:
Clinically, sympathetic blocks (SB) have been used widely to relieve the symptoms of SMP or to differentiate between SMP and sympathetically independent pain. In order to an SB has a diagnostic value, it requires the successful disturbance of the sympathetic activity for a proper duration of time.

For the diagnosis of SMP using an SB, it is essential achieving complete interruption of the sympathetic activity while preserving the sensory and motor function. The sympathetic trunk at lumbar region runs on the anterolateral surface of the vertebral column from L1 to L4 levels, and deep to the medial aspect of the psoas major muscle. Therefore, the investigators can hardly find epidural contrast spread during lumbar SB due to an anterior location of lumbar sympathetic ganglion to the lateral vertebral body. However, frequent psoas muscle injection can be encountered due to a close proximity of lumbar sympathetic ganglion.

In contrast to lumbar sympathetic ganglion, the thoracic sympathetic ganglion is not separated from somatic nerves by muscles and connective tissue. Moreover, the upper thoracic ganglion runs on the posterior surface of vertebral column with close proximity to adjacent epidural region.

This difference of thoracic sympathetic ganglion leads to a frequent epidural and intercostal spread if the investigators perform thoracic SB. Such spread to epidural and intercostal space lowers the diagnostic value of thoracic SB. In addition, serious adverse outcome can be encountered if neurolytic agent is injected into epidural or intercostal space for the purpose of thoracic sympathectomy. Considering the diagnostic value and safety of thoracic SB, evaluation of actual incidence of occurrence of intercostal and epidural spread is important.

ELIGIBILITY:
Inclusion Criteria:

* complex regional pain syndrome
* lymphedema after breast cancer surgery

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe unilateral arm pain or edema which is intractable to conservative therapy
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-06-23 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
incidence of intercostal spread | 60 seconds after the completion of thoracic sympathetic ganglion block. 60 seconds means the time when the outcome was measured after thoracic sympathetic ganglion block
  intercostal spread which appears at fluorosopic view after contrast medium injection
incidence of epidural spread | 60 seconds after the completion of thoracic sympathetic ganglion block. 60 seconds means the time when the outcome was measured after thoracic sympathetic ganglion block
  epidural spread which appears at fluorosopic view after contrast medium injection

SECONDARY OUTCOMES:
degree of finger tip skin temperature increase | 5, 10, 15, 20 minutes after the completion of the intervention 5, 10, 15, 20 minutes mean the time that the outcome was measured after performing the intervention
  Skin temperature measurement which is observed after successful sympathetic block

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (2):
- South Korea (2):
  - Hong ji HEE, Daegu
  - Ji Hee Hong, Daegu

IPD SHARING:
Plan to Share IPD: No